CLINICAL TRIAL: NCT04635215
Title: Observational Study of the Quality of Life of Patients With New Stoma Formation and Users of a Stoma Appliance From the SenSura Mio Range With Bodyfit® Technology
Brief Title: Observational Study of the Quality of Life of New Ostomates Using SenSura Mio Appliances With BodyFit Technology
Acronym: QoLMio
Status: Completed | Type: Observational
Sponsor: Laboratoires Coloplast S.A.S (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-A03232-53; 2018-A03232-53 (Other: ANSM (French competent authority)
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Ostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: There are not multiple groups in this study
  Interventions: Device: Sensura Mio Bodyfit technology ostomy pouches

INTERVENTIONS:
Device: Sensura Mio Bodyfit technology ostomy pouches — The use of medical devices, the ostomy pouches from Sensura Mio Bodyfit technology range, will be studied from inclusion visit (less than one month after the beginning of use) and during 3 months.

SUMMARY:
An ostomy is defined by the connection of a viscera to the skin, outside its natural location, by diversion from the digestive or urinary tract. The bodily injury, i.e. the creation of a stoma, has familiar, social and professional consequences. Personalized care, with the help of an ostomy nurse, is essential to accompany the ostomy patient in the changes of his or her life habits. In addition, the progress made in the various appliances, pouching and irrigation systems, contribute to improving the quality of life of these people.

In this context of adapted support, COLOPLAST has developed a range of ostomy pouches, the SenSura Mio BodyFit® technology range, for digestive or urinary stomas. The diversity of the devices makes it possible to find the most suitable combination to adapt to the morphology thanks to an elastic adhesive for a secure fit to individual body shape, and the textile materials used make it possible to optimize wearing comfort.

The aim of this study is to evaluate the quality of life of patients with recent ostomies with one of COLOPLAST's SenSura Mio devices at three months after discharge from the hospital. The condition of the skin around the stoma and the level of satisfaction of the patients will also be evaluated. Finally, the results obtained aim to identify factors predictive of a better quality of life in order to improve management.

DETAILED DESCRIPTION:
Today, there are about 80,000 people with ostomies in France and 19,000 ostomies are created each year.

An ostomy is defined by a viscera reaching the skin, outside its natural location, by diversion of the digestive (enterostomy) or urinary (ureterostomy) tract. Digestive ostomies are temporary or permanent palliative surgeries that consist of connecting a segment of the healthy digestive tract to the surface of the skin, either downstream or upstream of a lesion. There are several reasons for this type of stoma: following colorectal cancer or IBD (chronic inflammatory bowel disease), or to decompress and drain the digestive tract in occlusion, or to protect a digestive anastomosis by temporarily diverting the intestinal flow. Urinary ostomies are usually performed following bladder cancer or neurogenic bladder that has resulted in the removal of the bladderr. The urinary tract is then diverted to allow the evacuation of urine into an artificial pouch.

The bodily injury, the creation of a stoma, can have serious familiar, social and professional repercussions. An early follow-up from the preoperative phase and long-term technical and psychological support promote an adaptation of quality. Helping the patient to live well with his disability is a complex task that mobilizes the skills of a multidisciplinary team of caregivers. Mastery of surgical techniques for the creation of ostomies and close collaboration between the surgeon and the stoma therapist are essential for the personalized care of ostomy patients.

Advances in various devices, bag systems and irrigation systems are concrete means that contribute greatly to improving the patient's quality of life. In this context of technological advances, COLOPLAST has developed a range of devices for incontinent digestive and urinary stomas, SenSura Mio Technology BodyFit®. This range of pouches adapts to peristomal morphology and body movements due to an elastic adhesive for a secure fit to individual body shapes. In addition, the pouches are designed to remain discreet and maximize wearing comfort due to a neutral-grey color water-repellent textile material, invisible even under white clothing, and a full-circle prefilter to differ filter saturation for proven reduction of ballooning.

The objective of this study is to evaluate the use of SenSura Mio products in real-life conditions in patients with recent ostomies. For this purpose, we will use the Stoma-QoL specific quality of life scale, as well as the Peristomal Skin Condition Rating Scale (DET Score).

The Stoma-QoL tool was developed and validated specifically for ostomy patients in 2005 at the initiative of COLOPLAST and in close collaboration with international experts, with the aim of evaluating the impact of ostomy related concerns on the quality of life of ostomy patients on the one hand, and improving and facilitating their follow-up on the other hand. Potential items were formulated based on the results of a series of semi-structured interviews conducted with 169 adult subjects who had ostomies for a long time. The process resulted in a preliminary version of 37 items, administered repeatedly to 182 subjects with an ileostomy or colostomy. A psychometric selection of the items was performed using a Rasch model. The Stoma-QOL questionnaire has in its most refined version 20 questions covering 4 domains, not scored independently: sleep, intimate relationships, relationships with family and close friends, and social relationships with other people. This 20-item version has been validated internationally in ileo- or colostomized patients. On average, the value of the overall Stoma-QoL score was 58.5 with the lowest mean value (53.8) observed in France and the highest mean value (62.6) in Denmark. Stoma-QoL can be offered to ostomy patients who have already lived at least 1 month with their stoma and appliance.

The DET Score -also known as the Ostomy Skin Tool- is a measurement tool for assessing the extent and severity of peristomal skin problems. It was developed by Martins et al in 2008, at the initiative of COLOPLAST and in close collaboration with international experts, with the intention of improving the monitoring of peristomal skin conditions in ostomy patients and optimizing communication between healthcare professionals. The DET Score is divided into three areas: Discoloration (D), Erosion (E) and Tissue Proliferation (T). For each area, a maximum of 5 points can be awarded, 3 for the affected area and 2 for severity. The scores for each domain should be based solely on observations of each subject's skin, not on past experience. Photographs of problem skin are included in this rating scale and can be used as a guide for scoring severity. Once the score for each domain has been assessed, a total score is calculated by adding the numbers. A score of 0 represents normal skin while a score of 15 represents maximum skin severity around the stoma. The DET Score was validated in 2011 18: it is now widely used and has been translated into several languages. Skin problems are considered mild if DET Score ≤ 4; moderate if DET Score < 7; severe if DET Score ≥ 7. The mean value observed in an international study of more than 3,000 ostomy patients was 2.5 (± 2.8).

The objectives of the present study are multiple: to evaluate the quality of life of patients with recent ostomies using SenSura Mio appliances during the first three months following hospital discharge, to evaluate the condition of the peristomal skin during this same period and to look for factors predictive of a better quality of life. The data collected in this study will help to better document the factors influencing the quality of life of French patients with recent ostomies and the value of using the new SenSura Mio appliances. This study will also provide a better understanding of the incidence of skin problems in the early follow-up phase (first three months) and the main corrective actions taken by the ostomy nurses.

The QoL Mio study population will be composed of adults with recent ostomies (stoma preparation < 1 month), with liquid effluent (right colostomy, ileostomy, jejunostomy or urostomy), for whom healthcare professionals have recommended the use of SenSura Mio devices for ostomy care as part of the routine care. Because liquid effluents can seep under the adhesive on the skin, this population (ostomy with liquid effluents) has a higher risk of peristomal skin damage with irritant dermatitis by contact with corrosive effluents. The BodyFit technology (conforms to folds and irregularities of the skin) of SenSura Mio devices appears to be particularly suitable in this population to preserve the integrity of the peristomal skin.

ELIGIBILITY:
Inclusion Criteria

* Male or female aged over 18 year old
* Subject who signed the consent form
* Subject affiliated to a social security scheme or entitled to a social security benefit
* Subject with an ostomy less than one month old, with an expected stoma duration > 3 months
* Subject presenting an enterostomy with liquid effluents (right colostomy, ileostomy, jejunostomy) or a urostomy, user of a high flow or drainable pouch (Uro)
* Subjects for which the healthcare professional decided to use the SenSura Mio Technology BodyFit™ as the first permanent ostomy appliance after surgery as part of the care routines
* Subject educated in ostomy care and who manages it himself in an autonomous or assisted manner.

Exclusion criteria

* Vulnerable subject with regard to the regulations in force
* Pregnant, parturient or breastfeeding woman ;
* Subject deprived of liberty by judicial, medical or administrative decision;
* Minor subject;
* Subject legally protected or unable to express consent;
* Subject not affiliated or not benefiting from a social security system;
* Subject falling into several of the above categories;
* Subject who refused to participate in the study; and
* Subject participating in other research or clinical studies
* Subject for which stoma closure is scheduled before the end of the study
* A subject who, according to the investigator, has cognitive problems that prevent him or her from answering a questionnaire or for whom evaluation could be problematic.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The QoL Mio study population will consist of adults with recent ostomies (< 1 month after stoma creation) for whom healthcare professionals have recommended the use of SenSura Mio ostomy care devices as part of care routines.
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Stoma QoL score at 3 months | The primary outcome will be measured at 3 months
  The Stoma-QOL questionnaire has 20 questions covering 4 domains,: sleep, intimate relationships, relationships with family and close friends, and social relationships with other people.
  For each question, the answer ranges from 1 (always) to 4 (never). The points obtained for each of the 20 questions are added together to obtain an overall score. This raw summary score per patient in the 20-80 range will be converted into a final "0-100 score" where 0 indicates the worst Quality of Life and 100 the best Quality of Life. A table is available for converting raw scores into final scores.

SECONDARY OUTCOMES:
Stoma QoL score at 1 and 2 months | At 1 and 2 months
  The Stoma-QOL questionnaire has 20 questions covering 4 domains,: sleep, intimate relationships, relationships with family and close friends, and social relationships with other people.
  For each question, the answer ranges from 1 (always) to 4 (never). The points obtained for each of the 20 questions are added together to obtain an overall score. This raw summary score per patient in the 20-80 range will be converted into a final "0-100 score" where 0 indicates the worst Quality of Life and 100 the best Quality of Life. A table is available for converting raw scores into final scores.
DET Score | At 1, 2 and 3 months
  The DET Score is divided into three areas: Discoloration (D), Erosion (E) and Tissue Proliferation (T). For each area, a maximum of 5 points can be awarded, 3 for the affected area and 2 for severity. The scores for each domain should be based solely on observations of each subject's skin, not on past experience. Photographs of problem skin are included in this rating scale and can be used as a guide for scoring severity. Once the score for each domain has been assessed, a total score is calculated by adding the numbers. A score of 0 represents normal skin while a score of 15 represents maximum skin severity around the stoma.
Patient satisfaction | 3 months
  Patient satisfaction will be evaluated using a visual scale with a score comprised between 0 and 10. A score of 0 (lower value) means insatisfaction and a score of 10 (maximum) means total satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Meurette, MD, Principal Investigator — Nantes University Hospital
Locations (77):
- France (77):
  - Centre Hospitalier Du Pays D'Aix, Aix-en-Provence
  - Hotel Dieu, Angers
  - Centre Hospitalier d'Arras, Arras
  - Hopital de Mercy, Ars-Laquenexy
  - Centre Hospitalier Henri Mondor, Aurillac
  - Ch Henri Duffaut, Avignon
  - Clinique Belharra, Bayonne
  - Centre Hospitalier de Beauvais, Beauvais
  - Hopital Jean Minjoz, Besançon
  - Hopital La Cavale Blanche, Brest
  - Hopital Cote de Nacre, Caen
  - Centre Hospitalier de Douai, Cambrai
  - Hopital Du Pays D Autan, Castres
  - Hopital Manchester, Charleville-Mézières
  - Centre Hospitalier General, Châteauroux
  - Centre Hospitalier Du Cotentin Site de Cherbourg, Cherbourg Octeville
  - Hopital Beaujon, Clichy
  - Hopital Sud Francilien, Corbeil-Essonnes
  - Centre Georges François Leclerc, Dijon
  - Clinique Claude Bernard, Ermont
  - Cabinet infirmier, Étrelles
  - Centre Hospitalier Intercommunal Eure Seine, Évreux
  - Cabinet Infirmier, Flins-sur-Seine
  - Hopital Nord Ouest, Gleizé
  - Centre Hospitalier de Gonesse, Gonesse
  - Hopital Saint Louis, La Rochelle
  - Hopital La Source, La Source
  - Hopital Prive de L Estuaire, Le Havre
  - Pole Sante Sud, Le Mans
  - Centre Hospitalier Du Dr Schaffner, Lens
  - Hopital Robert Boulin, Libourne
  - Hopital Dupuytren, Limoges
  - Hopital Saint Philibert, Lomme
  - Hopital Nord, Marseille
  - Hopital Alphonse Laverand, Marseille
  - Hopital de La Conception, Marseille
  - Polyclinique Du Val de Saone, Mâcon
  - Centre Hospitalier Annecy Genevois Site Annecy, Metz-Tessy
  - Hopital Lapeyronie, Montpellier
  - Clinique St Augustin, Nantes
  - CHU Hôtel-Dieu, Nantes
  - Centre Hospitalier Georges Renon, Niort
  - Hopital Caremeau, Nîmes
  - Centre Hospitalier de Guingamp, Pabu
  - Hopital Saint Louis, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Cochin, Paris
  - Hopital Bichat Claude Bernard, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Tenon, Paris
  - Centre Hospitalier Francois Mitterand, Pau
  - Hopital Saint Jean, Perpignan
  - Clinique Mutualiste de Pessac, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire La Miletrie, Poitiers
  - Hopital Pontchaillou, Rennes
  - Centre Hospitalier de Rochefort, Rochefort
  - Hopital Charles Nicolle, Rouen
  - Hopital Yves Le Foll, Saint-Brieuc
  - Centre Hospitalier St Charles, Saint-Dié
  - Cabinet infirmier, Saint-Hilaire-de-Riez
  - Hopital Nord, Saint-Priest-en-Jarez
  - Les Hopitaux Du Mont Blanc, Sallanches
  - Centre Hospitalier de Salon de Provence, Salon-de-Provence
  - Centre Hospitalier de Seclin/Carvin, Seclin
  - Hopital Civil, Strasbourg
  - Hopital Hautepierre, Strasbourg
  - Centre Hospitalier de La Gespe, Tarbes
  - Hopitaux Du Leman Site Thonon, Thonon-les-Bains
  - Hopital Sainte Musse, Toulon
  - Hopital Rangueil, Toulouse
  - Hopital Des Hauts Clos, Troyes
  - Centre Hospitalier General, Valence
  - Polyclinique Vauban, Valenciennes
  - Centre Hospitalier de Valenciennes, Valenciennes
  - Hopitaux de Brabois, Vandœuvre-lès-Nancy
  - Hopital Robert Schuman, Vantoux

IPD SHARING:
Plan to Share IPD: No